CLINICAL TRIAL: NCT04455230
Title: A Multicenter, Long-term, Follow-up Study to Investigate the Safety and Durability of Response Following Dosing of an Adeno-associated Viral Vector (FLT190) in Subjects With Fabry Disease
Brief Title: A Long Term Follow-Up Study of Fabry Disease Subjects Treated With FLT190
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spur Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FLT190-02
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Fabry Disease; Lysosomal Storage Diseases
Keywords: Gene Therapy
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases

STUDY DESIGN:
Intervention Model Description: A Multicenter, Long-term, Follow-up Study to Investigate the Safety and Durability of Response Following Dosing of an Adeno-associated Viral Vector (FLT190) in Subjects with Fabry Disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants who have received gene therapy vector (FLT190) (Experimental)
  Interventions: Genetic: FLT190

INTERVENTIONS:
Genetic: FLT190 — FLT190 is a recombinant adeno-associated viral (AAV) vector (AAVS3) containing the human αGLA gene as a single stranded (ss) deoxyribonucleic acid (DNA).

SUMMARY:
Fabry disease is a rare, X-linked inborn error of glycosphingolipid metabolism caused by an abnormal gene encoding the α-galactosidase A (αGLA) enzyme. The αGLA enzyme is ubiquitously expressed throughout the body and is responsible for the breakdown of glycosphingolipids, deficiency of which results in the accumulation of specific glycosphingolipids that are associated with the pathophysiology of the disease. Current treatment for Fabry disease is limited to the symptomatic management of pain, conventional management of complications, and methods to increase the availability of functional αGLA.

This clinical study aims to investigate the long-term safety and durability of αGLA in patients who have been dosed with a new gene therapy product (FLT190) in earlier clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have previously received FLT190
* Provision of full informed consent and able to comply with all requirements of the study including long-term follow-up for 60 months (5 years) post-treatment.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Safety endpoint will be assessed by the reporting of adverse events (AEs) according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. | Entry to 5 years post dosing

CONTACTS AND LOCATIONS:
Locations (2):
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- Royal Free London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No